CLINICAL TRIAL: NCT00437073
Title: Study EGF107671 - a Phase II Study of Lapatinib Plus Topotecan or Lapatinib Plus Capecitabine in the Treatment of Recurrent Brain Metastases From ErbB2-Positive Breast Cancer Following Cranial Radiotherapy
Brief Title: Brain Metastases In ErbB2-Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lapatinib-topotecan arm enrollment closed early per protocol amendment 2. Then enrollment into remaining arm terminated due to operational issues.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107671
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2012-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Neoplasms, Breast
Keywords: brain metastases; ErbB2; lapatinib; Breast Cancer; HYCAMTIN; topotecan; capecitabine; metastatic breast cancer; TYKERB; XELODA
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Capecitabine; Topotecan; Lapatinib

ARMS (2):
- lapatinib plus capecitabine (Experimental): A total of 55 isubjects will be enrolled into this arm. Subjects with progression of CNS and/or non-CNS disease will be considered progressors. At the time of radiographically-documented CNS and/or non-CNS disease progression, a subject randomized to this arm will be allowed to cross over to the alternative arm.
  Interventions: Drug: capecitabine; Drug: lapatinib
- lapatinib + topotecan (Experimental): A total of 55 isubjects will be enrolled into this arm. Subjects with progression of CNS and/or non-CNS disease will be considered progressors. At the time of radiographically-documented CNS and/or non-CNS disease progression, a subject randomized to this arm will be allowed to cross over to the alternative arm.
  Interventions: Drug: topotecan; Drug: lapatinib

INTERVENTIONS:
Drug: capecitabine — capecitabine 2000mg/m2/day orally, Days 1-14, every 21 days
  Other Names: Xeloda
  Arms: lapatinib plus capecitabine
Drug: topotecan — topotecan intravenous (IV, in the vien) 3.2mg/m2 Days 1, 8 and 15; every 28 days
  Other Names: Hycamtin
  Arms: lapatinib + topotecan
Drug: lapatinib — lapatinib administered 1250mg once daily orally
  Other Names: Tykerb/Tyverb

SUMMARY:
This study is for patients with ErbB2 overexpressing breast cancer that has spread to the brain and is still progressing there even after radiation treatment using WBRT (whole brain radiotherapy) or SRS (stereotactic radiosurgery) to the brain. The study will determine how safe and effective lapatinib is when given in combination with capecitabine to treat patients with ErbB2 overexpressing breast cancer that has spread to the brain. Lapatinib is an oral drug that will be taken every day. Tests for safety and efficacy will be performed regularly during the course of the study.

ELIGIBILITY:
Inclusion criteria:

Subjects eligible for enrollment in the study must meet all of the following criteria:

* Signed written informed consent;
* Females or males age ≥ 18 years old;
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1;
* Life expectancy of at least 12 weeks;
* Subjects must have histologically or cytologically confirmed invasive breast cancer, with Stage IV disease;
* ErbB2 overexpressing breast cancer, defined as 3+ staining by immunohistochemistry (IHC), or 2+ staining by IHC in conjunction with ErbB 2 gene amplification by FISH, or ErbB 2 gene amplification by FISH alone (in subjects whose tumor blocks were not assessed by IHC). Subjects with tumors that are 2+ by IHC but negative or borderline by FISH assay are ineligible. For subjects with a history of more than one primary breast cancer, each breast cancer must be ErbB2 overexpressing to be eligible;
* ErbB2 overexpressing breast cancer, defined as 3+ staining by immunohistochemistry (IHC), or 2+ staining by IHC in conjunction with ErbB2 gene amplification by FISH, or ErbB2 gene amplification by FISH alone (in subjects whose tumor blocks were not assessed by IHC). ErbB2 gene amplification is defined by: > 6 ErbB2 gene copies/nucleus for test systems without an internal control probe or an ErbB2/CEP 17 ratio of more than 2.2. Subjects with tumors that are 2+ by IHC but negative or borderline by FISH assay are ineligible. For subjects with a history of more than one primary breast cancer, each breast cancer must be ErbB2 overexpressing to be eligible;
* Prior treatment of brain metastases with WBRT and/or SRS;
* Unequivocal evidence of new and / or progressive lesions in the brain on an imaging study; Note: Subjects with progressive brain lesions are not required to meet RECIST criteria for CNS progression in order to be eligible for this study.
* Prior treatment with trastuzumab, either alone or in combination with chemotherapy is required. Trastuzumab will be discontinued at least 2 weeks prior to enrollment on study;
* Cardiac ejection fraction within institutional range of normal as measured by echocardiogram. Subjects who require cardiac medications (e.g. positive inotropic agents or afterload reducers) for normal ejection fraction are ineligible. MUGA scans will be accepted in cases where an echocardiogram cannot be performed or is inconclusive;
* At least 2 weeks since prior radiotherapy, last chemotherapy, immunotherapy, biologic therapy, or hormonal therapy for cancer, and sufficiently recovered or stabilized from side effects associated with prior therapy. Concurrent treatment with bisphosphonates is permitted;
* At least 3 weeks since major surgical procedures;
* Able to swallow and retain oral medications;
* Women of childbearing potential must have a negative serum pregnancy test at screening and must use an approved contraceptive method, if appropriate (for example, intrauterine device [IUD], birth control pills, or barrier device) beginning 2 weeks before the first dose of investigational product and for 28 days after the final dose of investigational product. Males able to father a child must practice adequate methods of birth control or practice complete abstinence from intercourse from the first dose of investigational treatment until one week after the final dose of investigational treatment.
* Subjects must complete all screening assessments as outlined in the protocol;
* Normal organ and marrow function as defined by these LABORATORY VALUES : ANC (absolute neutrophil count) ≥ 1.5 x 10^9/L; Hemoglobin ≥ 10 g/dL (after transfusion if needed); Platelets ≥ 100 x 10^9/L; Albumin ≥ 2.5 g/dL; Serum bilirubin ≤ 1.5x ULN unless due to Gilbert's syndrome; AST and ALT ≤ 5x ULN if documented liver metastases ≤ 3x ULN without liver metastases; Serum Creatinine ≤ 1.2 mg/dL or Calculated Creatinine Clearance1 ≥ 50 mL/min

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Subjects who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or who have unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment;
* Concurrent treatment with an investigational agent or participation in another treatment clinical trial;
* Prior therapy with a topoisomerase 1 inhibitor;
* Prior lapatinib therapy;
* Prior therapy with capecitabine;
* Known dihydropyrimidine dehydrogenase (DPD) deficiency;
* ECOG Performance Status 2 or greater;
* Subjects receiving concurrent chemotherapy, radiation therapy, immunotherapy, biologic therapy (including an ErbB1 and/or ErbB2 inhibitor), or hormonal therapy for treatment of their cancer. Hormone therapy for ovarian suppression which has been used for > 6 months, during which time there has been disease progression in the brain, is allowed. Concurrent treatment with bisphosphonates is allowed;
* Subjects with evidence of leptomeningeal carcinomatosis at screening;
* History of allergic reactions attributed to compounds of similar chemical composition (quinazolines) to lapatinib;
* History of allergic reactions attributed to compounds chemically related to capecitabine, fluorouracil or any excipients;
* Concurrent treatment with medications listed as Prohibited Medications;
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with active, uncontrolled ulcerative colitis are also excluded;
* History of immediate or delayed hypersensitivity reaction to gadolinium contrast agents, or other contraindication to gadolinium contrast;
* Other known contraindication to MRI, such as a cardiac pacemaker, implanted cardiac defibrillator, brain aneurysm clips, cochlear implant, ocular foreign body, or shrapnel;
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical or psychiatric disorder that would interfere with the subject's safety;
* Anticoagulant therapy (other than coumadin or aspirin as catheter prophylaxis) at study entry;
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent, unless a legally acceptable representative could provide informed consent (if in accord with the policies of the local Ethics Committee);
* Pre-existing severe cerebral vascular disease, such as stroke involving a major vessel, CNS vasculitis, or malignant hypertension;
* Active cardiac disease, defined as one or more of the following:
* History of uncontrolled or symptomatic angina
* History of arrhythmias requiring medications, or clinically significant
* Myocardial infarction < 6 months from study entry
* Uncontrolled or symptomatic congestive heart failure
* Ejection fraction below the institutional normal limit
* Any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient;
* Uncontrolled infection;
* Pregnant or lactating females;
* History of other malignancy, except for curatively treated basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix. Subjects with other malignancies who have been disease-free for at least 5 years are eligible.
* Have current active hepatic or biliary disease (with exception of subjects with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2009-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- United States (13):
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Sioux City, Iowa
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Dallas, Texas
- Austria (2):
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- GSK Investigational Site, Brussels, Belgium
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Québec, Quebec
- France (4):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Herblain
- Germany (4):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Bremen, City state Bremen
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Troisdorf, North Rhine-Westphalia
- Greece (2):
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Neo Faliro
- Israel (3):
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Zrifin
- Italy (2):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Perugia, Umbria
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Hospitalet de Llobregat, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Uppsala, Sweden

REFERENCES:
- [Background] Lin NU, Eierman W, Greil R, Campone M, Kaufman B, Steplewski K, Lane SR, Zembryki D, Rubin SD, Winer EP. Randomized phase II study of lapatinib plus capecitabine or lapatinib plus topotecan for patients with HER2-positive breast cancer brain metastases. J Neurooncol. 2011 Dec;105(3):613-20. doi: 10.1007/s11060-011-0629-y. Epub 2011 Jun 26. PMID 21706359

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib Plus Capecitabine: Participants received a daily dose of 5 tablets of lapatinib (1250 milligrams [mg]) at approximately the same time every day, either 1 hour (or more) before breakfast or 1 hour (or more) after breakfast. Participants also received capecitabine 2000 mg per meters squared (mg/m^2) per day, divided and administered orally twice daily, 12 hours apart, for 14 days, every 21 days. Capecitabine was taken with food or within 30 minutes after a breakfast meal with approximately 200 milliliters (ml) of water.
- Lapatinib Plus Topotecan: Participants received a daily dose of 5 tablets of lapatinib (1250 milligrams [mg]) at approximately the same time every day, either 1 hour (or more) before breakfast or 1 hour (or more) after breakfast. Participants also received an intravenous (IV) infusion of topotecan 3.2 mg/m^2 over the course of at least 30 minutes on Days 1, 8, and 15 (+/- 2 days) of a 28-day treatment cycle.
Period: Overall Study
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Started | 13 | 9
Completed | 12 | 8
Not Completed | 1 | 1
Not completed — Sponsor Terminated Study | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (9.29) | 54.6 (10.54) | 51.5 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Central Nervous System (CNS) Objective Response (OR)
Description: CNS OR is defined as the number of participants with either a complete response (CR) or partial response (PR) as assessed by volumetric analysis of brain magnetic resonance imaging (MRI) and Response Evaluation Criteria In Solid Tumors (RECIST). CR: complete resolution of all evaluable and non-evaluable brain metastases; PR: =>50% reduction in the volumetric sum of all evaluable brain metastases compared to baseline.
Time Frame: From the start of treatment until disease progression, death, or discontinuation from the study, up to a maximum of Week 88
Population: Modified Intent-to-Treat (mITT) Population: all participants who had at least one evaluable CNS target lesion at baseline and who had received at least two doses of lapatinib medication
Measure: Number; unit: participants
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 13 | 9
participants | 5 | 0
Statistical Analysis 1: Comparison: Lapatinib Plus Capecitabine; Test type: Superiority or Other; percentage of participants = 38, 95% CI 2-sided [13.9 to 68.4] — The estimated value indicates the percentage of participants with CNS OR in the Lapatinib plus Capecitabine treatment arm

2. Primary Outcome: Number of Participants With the Indicated CNS Responses
Description: CNS responses were assessed by volumetric (V) analysis of brain MRI and RECIST. CR: complete resolution of all evaluable and non-evaluable brain metastases (BMs). PR: =>50% reduction in the V sum of all evaluable BMs compared to baseline. A response of "Other" was used for participants who discontinued the study prior to the first efficacy assessment. Stable Disease (SD): disease that does not meet CR, PR, or CNS progression criteria. Progressive disease (PD): a requirement for a new steroid or an increasing steroid dose for the treatment of worsening neurological signs/symptoms due to BMs.
Time Frame: as for outcome 1
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 13 | 9
participants
  Complete response | 0 | 0
  Partial response | 5 | 0
  Stable Disease | 6 | 3
  Progressive Disease | 2 | 1
  Unknown | 0 | 3
  Other | 0 | 2

3. Secondary Outcome: Duration of CNS Objective Response (Defined as the Time From the First Documented Evidence of CNS PR or CR Until the First Documented Sign of Disease Progression or Death, if Sooner)
Description: CNS OR is defined as the number of participants with either a CR or PR as assessed by volumetric analysis of brain MRI and RECIST. CR: complete resolution of all evaluable and non-evaluable brain metastases; PR: =>50% reduction in the volumetric sum of all evaluable brain metastases compared to baseline. This study was closed before full enrollment was achieved; thus, predefined secondary efficacy endpoints were not assessed because there were not enough participants enrolled in the study to provide statistically valid analyses.
Time Frame: as for outcome 1
Population: mITT Population
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical benefit is defined as CR (complete resolution of all evaluable and non-evaluable brain metastases), PR (=>50% reduction in the volumetric sum of all evaluable brain metastases compared to baseline), or stable disease (disease that does not meet CR, PR, or CNS progression criteria) for at least 6 months. This study was closed before full enrollment was achieved; thus, predefined secondary efficacy endpoints were not assessed because there were not enough participants enrolled in the study to provide statistically valid analyses.
Time Frame: as for outcome 1
Population: mITT Population
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants (Par.) With Objective Response by RECIST in Non-CNS Disease
Description: Non-CNS disease (for par. with measurable baseline non-CNS disease) OR is defined as the number of par. with either a CR or PR as assessed by computed tomography (CT) or MRI scan and RECIST. CR: disappearance of all target lesions; PR: at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. This study was closed before full enrollment was achieved; thus, predefined secondary efficacy endpoints were not assessed because there were not enough par. enrolled in the study to provide statistically valid analyses.
Time Frame: as for outcome 1
Population: mITT Population
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to CNS Objective Response (Defined as the Time From the Start of Treatment Until the First Documented Evidence of Partial or Complete Tumor Response [Whichever Status is Recorded First])
Description: as for outcome 3
Time Frame: as for outcome 1
Population: mITT Population
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With the Indicated Site of Initial Disease Progression
Description: The site of initial disease will be determined by taking the earliest date of known progression and assigning the appropriate category (CNS or non-CNS) based on the source of the earliest date. This study was closed before full enrollment was achieved; thus, predefined secondary efficacy endpoints were not assessed because there were not enough participants enrolled in the study to provide statistically valid analyses.
Time Frame: as for outcome 1
Population: mITT Population
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from the start of treatment until the first documented sign of disease progression at any site or death due to any cause, if sooner. This study was closed before full enrollment was achieved; thus, predefined secondary efficacy endpoints were not assessed because there were not enough participants enrolled in the study to provide statistically valid analyses.
Time Frame: as for outcome 1
Population: mITT Population
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the start of treatment until death due to any cause. This study was closed before full enrollment was achieved; thus, predefined secondary efficacy endpoints were not assessed because there were not enough participants enrolled in the study to provide statistically valid analyses.
Time Frame: as for outcome 1
Population: mITT Population
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percentage of Participants With Baseline Tumor-related (TR) Neurological Signs and Symptoms (NSS), Who Experienced Improvement in NSS as Measured by the Neurological Examination Worksheet (NEW)
Description: TR NSS was to be recorded by the Investigator on the NEW, using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE V3.0). Improvement was to be defined as a decrease of 1 or more CTCAE grades from baseline of any TR NSS. This study was closed before full enrollment was achieved; thus, predefined secondary efficacy endpoints were not assessed because there were not enough participants enrolled in the study to provide statistically valid analyses.
Time Frame: as for outcome 1
Population: mITT Population
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percentage of Participants With Disease Stabilization for 6 Months or More
Description: The percentage participants with disease stabiliztion for 6 months or more were defined as those treated participants with a best CNS objective response of SD whose disease stabilization lasted 6 months or more from the start of treatment. This study was closed before full enrollment was achieved; thus, predefined secondary efficacy endpoints were not assessed because there were not enough participants enrolled in the study to provide statistically valid analyses.
Time Frame: as for outcome 1
Population: mITT Population
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants With a >=20% Volumetric Reduction in CNS Lesions
Description: The percentage of participants with a >=20% volumetric reduction in CNS lesions was defined as the percentage of treated participants achieving at least a 20% volumetric reduction in CNS lesions relative to baseline. This study was closed before full enrollment was achieved; thus, predefined secondary efficacy endpoints were not assessed because there were not enough participants enrolled in the study to provide statistically valid analyses.
Time Frame: Baseline; from the start of treatment until disease progression, death, or discontinuation from the study, up to a maximum of Week 88
Population: mITT Population
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All serious and non-serious on-therapy adverse events, defined as occurring from the first dose of investigational product until five days after the last dose (up to Week 37) were recorded, regardless of whether or not they were considered drug related.
Description: Serious and non-serious adverse events were collected in members of the ITT Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Topotecan
Serious Adverse Events (participants affected / at risk) | 6/13 | 5/9
Other Adverse Events (participants affected / at risk) | 13/13 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Plus Capecitabine (N=13) | Lapatinib Plus Topotecan (N=9)
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Plus Capecitabine (N=13) | Lapatinib Plus Topotecan (N=9)
Diarrhoea (Gastrointestinal disorders) | 11 | 8
Nausea (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 8 | 5
Oedema peripheral (General disorders) | 5 | 0
Mucosal inflammation (General disorders) | 4 | 0
Asthenia (General disorders) | 1 | 1
Oedema (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Facial pain (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 3
Dizziness (Nervous system disorders) | 3 | 2
Dysgeusia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Muscle contraction involuntary (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 5
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 2
Weight decreased (Investigations) | 1 | 1
Activated partial thromboplastin time shortened (Investigations) | 0 | 1
Alanine aminotransferase (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin (Investigations) | 0 | 1
Blood glucose abnormal (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood phosphorus decreased (Investigations) | 1 | 0
Protein total abnormal (Investigations) | 1 | 0
Prothrombin time abnormal (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Depressed mood (Psychiatric disorders) | 2 | 0
Hot flush (Vascular disorders) | 1 | 1
Infection (Infections and infestations) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Abscess (Infections and infestations) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral fungal infection (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
White blood cell count decreased (Blood and lymphatic system disorders) | 0 | 1
Disorientation (Nervous system disorders) | 1 | 0
Dry eyes (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.